CLINICAL TRIAL: NCT03009084
Title: Nephrocare: Multidisciplinary Care for Patients With Chronic Kidney Disease: an Increase of Patient Empowerment and Self-management by Using Interactive and Communication Tools and Nursing Interventions.
Brief Title: Multidisciplinary Care for Patients With Chronic Kidney Disease to Increase Their Self-management.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Kathleen Claes, Prof. Dr., Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: S57777
Record Dates: First submitted 2015-04-11; First posted 2017-01-04 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (Experimental): Lifestyle counseling of modifiable risk factors of chronic kidney disease: telemonitoring of blood pressure, counseling for smoking cessation, losing weight and increasing the physical activity.
  Interventions: Behavioral: Lifestyle counseling
- Control group (No Intervention): Usual care.

INTERVENTIONS:
Behavioral: Lifestyle counseling — Lifestyle counseling of modifiable risk factors of chronic kidney disease: telemonitoring of blood pressure, counseling for smoking cessation, losing weight and increasing the physical activity.
  Arms: Intervention group

SUMMARY:
The purpose of this study is to investigate the communication and data sharing between the primary care physician and the nephrologist about patients with chronic kidney disease. Also therapeutic interventions that change behavior and telemonitoring of the blood pressure will be explored and compared to the usual care. The most important aim of this study is to improve the quality of care for the patient with chronic kidney disease in cooperation with the primary care physician and the nephrologist.

DETAILED DESCRIPTION:
Through questionnaires with primary care physicians, nephrologists from the University Hospitals of Leuven and patients with chronic kidney disease, the problems will be known.

After the exploration there will be an intervention with patients who meet the in- and exclusion criteria. Around 150-200 patients will be included with a 1:2 randomisation in the control and intervention group. The relevant clinical data and the factors of lifestyle will be questioned at the baseline.

The intervention group will receive individualized therapy by a nurse, for example to quit smoking, to eat healthier and to do more physical activities. This therapy is based on the most important risk factors and will be determined before the start of the therapy. Further on, these patients will also be motivated to take their blood pressure more frequently by using a telemonitoring system.

ELIGIBILITY:
Inclusion Criteria:

* Predialysis, hemodialysis, peritoneal dialysis, transplantation
* Included in the care program of chronic kidney diseases
* Dutch-speaking
* Signed and approved informed consent

Exclusion Criteria:

* No Dutch-speaking
* Impaired cognitive condition or medically unstable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2015-09-17 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
BMI change | one year
  BMI change in kg/m²
smoking cessation | one year
  percentage of smoking cessation.
change in Estimated Glomerular Filtration Rate (eGFR) | one year
  Estimated Glomerular Filtration Rate (eGFR) in mL/min/1.73m²
lipid control | one year
  LDL in mmol/l
blood pressure under control | one year
  percentage of patients with blood pressure within target limits

SECONDARY OUTCOMES:
Communication between primary care physicians and the nephrologists. | 6 months
  Improved communication between primary care physicians and nephrologists measured by a questionnaire.
Relevant clinical data: systolic and diastolic blood pressure | one year
  Improved or stable clinical data that are taken at the consultation of nephrology (systolic and diastolic blood pressure).

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Claes, Prof. Dr., Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided